CLINICAL TRIAL: NCT03340207
Title: Clinical Trial of PneumaGlide: A Novel Airway Device to Aid Endotracheal Intubations for Novice Intubators
Brief Title: Novel Airway Device to Aid Endotracheal Intubations
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: A longer time to establish the airway. potential safety issue, despite lacking no adverse event.
Sponsor: University at Buffalo (Other)
Responsible Party: Principal Investigator, Nader D Nader, Professor and Senior Vice Chair, University at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1092558
Record Dates: First submitted 2017-11-08; First posted 2017-11-13 (Actual); Results first posted 2022-10-14 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-09

CONDITIONS: Intubation Complication; Intubation;Difficult
Keywords: intubation; anesthesiology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Pneumaglide (Experimental): After induction of anesthesia Pneumaglide device will be placed in the mouth of the pneumaglide assigned patients.
  Interventions: Device: Pneumaglide
- non-pneumaglide (No Intervention): The patients in non-pneumaglide will not have Pneumaglide insertion prior to intubation.

INTERVENTIONS:
Device: Pneumaglide — The device is designed to facilitate intubation and reduce the time to intubation. It works with traditional glidescope to make the process of intubation easier. In this study patients scheduled for surgery and intubation, will be randomized to two groups. The intervention group will be intubated with the help of the pneumaglide. Yet, the other group will receive standard intubation. We aim to evaluate the efficacy of the Pneumaglide to improve the ease of intubation in unskilled clinicians and skilled clinicians during difficult and routine intubations
  Arms: Pneumaglide

SUMMARY:
Pneumaglide is a device designed to facilitate intubation. Patients who are undergoing a surgical procedure under general anesthesia and will require placement of endotracheal tube will be screened and upon fulfilling the inclusion criteria will be randomized to PneumaGlide group or non-PneumaGlide group. After induction of anesthesia PneumaGlide device will placed in the mouth of the Pneumaglide assigned subject. The time for intubation will be measured from the time that the laryngoscope is inserted into the mouth until the trachea is successfully intubated and compared between the groups. Oxygen saturation drop below 90% and also gastric secretion spillage will be compared between two groups as well.

DETAILED DESCRIPTION:
Patients who is undergoing a surgical procedure under general anesthesia and will require placement of endotracheal tube will be screened. If the patient meets the inclusion criteria and does not have any exclusion criteria, after an informed consent is obtained he or she will be randomized to Pneumaglide group or non-Pneumaglide group . Patients characteristics, anthropometric data and comorbid conditions wil be questioned and collected into data collection tool forms. Airway difficulty will be assessed by the range of motion for atlanto axial joint (head flexion and extension), temporomandibular joint (mouth opening), thyromental distance and mallampati classification for visualisation of uvula, tonsillar pillars and soft palate. After induction of anesthesia PneumaGlide device will placed in the mouth of the pneumaglide assigned subject. The patients in non-pneumaglide will not have Pneumaglide insertion. Laryngeal grading of the airway difficulty will be determined in both groups and the degree of difficulty will be graded from I-IV based on visibility of the vocal cords. The time will be measured using a an electronic timer from the time that the laryngoscope is inserted into the mouth until the trachea is successfully intubated. The spillage of of gastric contents will also be assessed by direct visualization at the time of intubation. Oxygen Saturation will be monitored throughout the case and any events with oxygen saturation levels < 90% will be recorded and compared in the two study arms. All Categorical variables will be analyzed using Fisher's exact test and the numerical values with normal distribution pattern will be analyzed with t-tests and expressed as mean ± standard deviation. Numerical variables in which the normality is rejected will be analyzed using non-parametric test Wilcox Sum Rank and will be expressed as median [Interquartile Range]. Upon completion of the surgery, two Likert-based questionaires will be filled out. One questionaire is completed by the person who performed intubation for the ease of use, and the level of comfort during its use. The second questionaire is handed to the patient at the time of their discharge from the Ambulatory Surgery Unit and will accompany a self addressed envelope. The patients will be asked for the presence of cough, shortness of breath, sore through, any unrecognized injury to the lip or mucosa of the mouth. The patients will be instructed to complete and mail their questionaire along with their mailing address.

ELIGIBILITY:
Inclusion Criteria:

* undergoing ambulatory surgery under general anesthesia

Exclusion Criteria:

* pregnant patients
* parturients with past 60 days,
* poorly controlled diabetic patient with neuropathy and HbA1c > 9.0%, *preexisting nausea and vomiting,
* intestinal obstruction
* acute alcohol toxicity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-10-15 (Actual); Primary Completion 2019-03-25 (Actual); Study Completion 2019-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nader D Nader, MD, PhD, Principal Investigator — University at Buffalo
Locations (1):
- Buffalo VA Medical Center, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make data available to others

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Requiring endotracheal intubation for general anesthesia
Pre-assignment Details: Group, age, BMI, Mallampathi class, Pre and post laryngeal grade of the airway, success and the number of attempts to intubate. As the main outcome variable, we collected the time it took to secure the airway. The occurrence of esophageal intubation, gastric aspiration, and injury to the oropharyngeal tissue was also documented.
Groups:
- Device: A total of 32 patients were randomized. 16 patients were randomized for Pneumoglide (PG).
- Control: the other 16 were assigned to the control group.
Period: Overall Study
Arm/Group | Device | Control
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Controls: 16 patients were randomized to the "No device" group
- Device: 16 patients were randomized to the "Pneumoglide" group
- Total: Total of all reporting groups
Arm/Group | Controls | Device | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants] — Age Category
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 13 | 15 | 28
    >=65 years | 3 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.6 (8.6) | 65.3 (7.8) | 66.7 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 16 | 16 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 2 | 3 | 5
  Unknown or Not Reported | 13 | 13 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 12 | 13 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 32
BMI [Mean (Standard Deviation); unit: kg/m^2] | 30.0 (7.6) | 32 (8.4) | 31 (7.5)
Mallampathi class [Number; unit: participants] — Number of the participants with Mallampati < Class 3 Mallampati class is used to assess the difficulty of the airway in a scale of 1-4. M1 stands for the easiest access while M4 stand for the most difficult airway.
  participants | 16 | 13 | 29
post laryngeal grade [Median (Inter-Quartile Range); unit: units on a scale] — The laryngeal view grades are as Grade 1: whole vocal cords are seen, but the epiglottis is not seen. Grade 2: larynx plus the posterior surface of epiglottis are seen. Grade 3: the anterior tip of the epiglottis is seen
  units on a scale | 2 [1 to 3] | 3 [1 to 3] | 2 [1 to 3]

OUTCOME MEASURES:

1. Primary Outcome: Time to Intubation
Description: After induction of anesthesia PneumaGlide device will be placed in the mouth of the pneumaglide assigned subject. The patients in non-pneumaglide will not have Pneumaglide insertion. Laryngeal grading of the airway difficulty will be determined in both groups and the degree of difficulty will be graded from I-IV based on visibility of the vocal cords. Grade I is full visibility of glottis, grade II is partial visibility of glottis, grade III is when only epiglottis seen, none of glottis seen, and finally grade IV is when neither glottis nor epiglottis seen. Accordingly higher values represent worse grade. The time will be measured using a an electronic timer from the time that the laryngoscope is inserted into the mouth until the trachea is successfully intubated.
Time Frame: During procedure
Population: time to intubate
Measure: Median (Inter-Quartile Range); unit: Seconds
Arm/Group | Pneumaglide | Non-pneumaglide
Number analyzed (Participants) | 16 | 16
Seconds | 56 [47 to 75] | 41 [37 to 48]

2. Secondary Outcome: Oxygen Saturation Drop
Description: Oxygen Saturation will be monitored throughout the case and any events with oxygen saturation levels < 90% will be recorded and compared in the two study arms.
Time Frame: during procedure
Population: pulseoxymetry
Measure: Count of Participants; unit: Participants
Groups:
- Control: 16 subjects were assigned to the control group.
- PneumaGlide: 16 subjects were randomised to this experimental group.
Arm/Group | Control | PneumaGlide
Number analyzed (Participants) | 16 | 16
Participants | 0 | 0

3. Secondary Outcome: Frequency of Lip/Dentition Injury
Description: frequency of lip/dentition injury will be monitored and compared
Time Frame: during procedure
Measure: Number; unit: participants
Arm/Group | Device | Control
Number analyzed (Participants) | 16 | 16
participants | 0 | 0

4. Secondary Outcome: Frequency of Ask for Help and Repeated Intubation Attempt
Description: Frequency of asking for help from seniors and repeated attempts for intubation will be recorded in each group
Time Frame: during procedure
Population: frequency
Measure: Count of Participants; unit: Participants
Groups:
- Device: 16 patients were randomized for Pneumoglide.
Arm/Group | Device | Control
Number analyzed (Participants) | 16 | 16
Participants | 3 | 0

5. Other Pre Specified Outcome: Adverse Event Reports by the Patients (Likert Scale)
Description: questionaire is handed to the patient at the time of their discharge from the Ambulatory Surgery Unit and will accompany a self addressed envelope. The patients will be asked for the presence of 1-cough, 2-shortness of breath, 3-sore through, 4-any unrecognized injury to the lip or mucosa of the mouth. Each answer is on a scale of 1-5 with 1representing minimal and 5 representing extremely severe complaint. Accordingly the score will be between 4-20. The patients will be instructed to complete and mail their questionaire along with their mailing address.
Time Frame: upon discharge from hospital up to two weeks
Population: This particular outcome measure reflects the number of the responders to the small questionnaire. While the initial number of the patients were 16 in each group, only 10 from the device group and 8 from the control group opted to respond and were included in the analysis.
Measure: Median (95% Confidence Interval); unit: total score on a scale 4-20
Groups:
- Device: 16 patients were randomized for Pneumoglide (PG).
- Control: 16 were assigned to the control group.
Arm/Group | Device | Control
Number analyzed (Participants) | 10 | 8
total score on a scale 4-20 | 5 [4 to 7] | 5 [5 to 8]

ADVERSE EVENTS:
Time Frame: Two weeks from the time of surgery
Description: lip injury, loss of airway, difficulty in intubation, gastric aspiration
Arm/Group | Device | Control
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-04-15): https://cdn.clinicaltrials.gov/large-docs/07/NCT03340207/Prot_SAP_ICF_000.pdf